CLINICAL TRIAL: NCT00395980
Title: Muscle Pressure in the Flank Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Responsible Party: Leslie Deane, MD, University of California, Irvine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2006-5106
Record Dates: First submitted 2006-11-02; First posted 2006-11-06 (Estimated); Last update posted 2008-12-12 (Estimated); Status verified 2008-12

CONDITIONS: Tissue Breakdown

INTERVENTIONS:
Device: surgical table pressure mat

SUMMARY:
Using healthy volunteers, participants will lay on an operating room table in various positions employed during kidney surgery. Using a pressure sensor mat, we hope to determine which areas of the body are subject to higher pressures. Using padding devices (foam, gel, water mattress)which are currently used in the operating room will be employed and measurements will be taken to determine which padding material and configurations is optimal to reduce the pressure to those body parts at risk for excessive pressure subject during laparoscopic surgery.

ELIGIBILITY:
Exclusion Criteria:

* Subjects with musculoskeletal disabilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-10; Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie A. Deane, MD, Principal Investigator — University of California, Irvine
Locations (1):
- University of California, Irvine Medical Center, Orange, California, United States